CLINICAL TRIAL: NCT05620940
Title: A PHASE 1, OPEN-LABEL, EXPLORATORY, FIXED-SEQUENCE, PHARMACOKINETIC SINGLE ASCENDING DOSE STUDY OF IVL3004 VERSUS VIVITROL® (NALTREXONE) LONG-ACTING INJECTABLE (LAI) AND IVL4002 IN HEALTHY SUBJECTS
Brief Title: A Clinical Trial to Assess Pharmacokinetic Profiles, Safety and Tolerability of IVL3004 and IVL4002 in Healthy Male Subjects.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Inventage Lab., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IVL3004-001
Record Dates: First submitted 2022-11-10; First posted 2022-11-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Opioid Dependence; Alcohol Dependence; Multiple Sclerosis
MeSH Terms: conditions — Opioid-Related Disorders; Alcoholism; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A Group 1 (Vivitrol Injection) (Active Comparator): Vivitrol, Single Dose, IM injection
  Interventions: Drug: Vivitrol Injectable Product
- Part A Group 2 (IVL3004 A mg) (Experimental): IM, Single Dose
  Interventions: Drug: IVL3004
- Part A Group 3 IVL3004 B mg) (Experimental): IM, Single Dose
  Interventions: Drug: IVL3004
- Part B Group 1 (IVL4002 Cmg) (Experimental): SC, Single Dose
  Interventions: Drug: IVL4002

INTERVENTIONS:
Drug: Vivitrol Injectable Product — Naltrexone Long-Acting Injection
  Arms: Part A Group 1 (Vivitrol Injection)
Drug: IVL3004 — Naltrexone Long-Acting Injection
  Arms: Part A Group 2 (IVL3004 A mg); Part A Group 3 IVL3004 B mg)
Drug: IVL4002 — Naltrexone Long-Acting Injection
  Arms: Part B Group 1 (IVL4002 Cmg)

SUMMARY:
A Clinical Trial to Assess Pharmacokinetic Profiles, Safety and Tolerability of IVL3004 and IVL4002 in Healthy Male Subjects.

DETAILED DESCRIPTION:
A Phase 1, Open-Label, Exploratory, Fixed-Sequence, Pharmacokinetic Single Acending Dose Study of IVL3004 Versus Vivitrol® (Naltrexone) Long-Acting Injectable(LAI) and IVL4002 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male, ≥18 and ≤55 years of age, non-smokers or occasional smokers (defined as smoking less than 10 cigarettes or nicotine equivalent per week, and willing to abstain from smoking during confinement at the clinical site).
2. BMI ≥18.0 and ≤32.0 kg/m2 and body weight ≥55.0 kg.
3. Healthy as defined by:

   1. The absence of clinically significant illness, infection, or medical/surgical procedure within 4 weeks prior to dosing or planned inpatient surgery (including dental surgery) or hospitalization during the study period.
   2. The absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological (including autoimmune), psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
4. Subjects who are not vasectomized for at least 3 months prior to dosing, and who are sexually active with a female partner of childbearing potential must be willing to use one of the following acceptable contraceptive methods from dosing and for 90 days after dosing:

   a. Simultaneous use of a male condom and, for the female partner, hormonal contraceptives used for at least 4 weeks or intrauterine device placed for at least 4 weeks prior to dosing.
5. Subjects who have had a vasectomy must be willing to use a condom until study exit.
6. Subjects who practice abstinence from sexual intercourse as a usual and preferred lifestyle.
7. Subjects must be willing not to donate sperm for 90 days after dosing.
8. Willing to undergo SC abdominal injection or IM ventral gluteal injection to allow for investigational drug administration.
9. Willing and able to provide written informed consent after the nature of the study has been explained and prior to the commencement of any protocol- specific study procedures.

Exclusion Criteria:

1. Any clinically significant abnormal finding at physical examination at screening or Day -1.
2. Clinically significant abnormal laboratory test results at screening or Day -1, or positive serology test results for human immunodeficiency virus (HIV), hepatitis B or hepatitis C virus at screening.
3. Is prone to skin rashes, irritation, or has a skin condition such as recurrent eczema that is likely to impact the injection site area or demonstrates any abnormal skin tissue in the proposed injection area, as determined by the Investigator.
4. Any history of malignancy or neoplastic disease.
5. History of significant allergic reactions (e.g., drug reaction, anaphylactic reaction, hypersensitivity, angioedema) to any drug, or to any excipient present in the formulations.
6. ALT, AST, or total bilirubin >1.5x upper limit of normal (ULN) at screening or Day -1.
7. Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2 as calculated by the 2021 Chronic Kidney Disease-Epidemiology (CKD-EPI) equation at screening or Day -1.
8. Clinically significant ECG abnormalities (QTc >450 ms or PR interval >220 ms) or vital sign abnormalities (systolic blood pressure <90 or >140 mmHg, diastolic blood pressure <40 or >90 mmHg, or heart rate <40 or >100 bpm) at screening or Day -1.
9. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 14 units of alcohol per week (1 unit = 375 mL of beer 3.5%, 100 mL of wine 13.5%, or 30 mL of spirit 40%), or positive alcohol test at screening or Day -1.
10. History of drug abuse within 1 year prior to screening or positive test for drugs of abuse (e.g., phencyclidine, opiates, benzodiazepines, barbiturates, amphetamines, methamphetamines, cocaine, and tetrahydrocannabinol) at screening or Day -1.
11. Presence of any underlying physical or psychological (e.g., depression) medical condition that, in the opinion of the Investigator, would make it unlikely that the participant will comply with the protocol or complete the study per protocol. Mild depression and anxiety that has been resolved at least 6 months prior to screening is accepted.
12. Use of medications for the timeframes specified below, with the exception of hormonal contraceptives and medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the PK profile of the study drug or subject safety:

    1. Depot injection or implant within 3 months prior to dosing;
    2. Strong CYP inhibitors or inducers within 30 days prior to dosing;
    3. Prescription medications within 14 days prior to dosing;
    4. Any vaccine, including COVID-19 vaccine, within 7 days prior to dosing;
    5. OTC medications (including topical and nasal formulations with active pharmaceutical ingredients) within 7 days prior to dosing, except for occasional use of acetaminophen/paracetamol (up to 2 g/day);
    6. Natural health products (including herbal remedies, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to dosing;
    7. Anesthetic agents within 24 hours prior to dosing.
    8. Anticoagulant medications from 15 days prior to dosing to 6 weeks post- dose.
13. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to dosing, administration of a biological product in the context of a clinical research study within 90 days prior to dosing, or concomitant participation in an investigational study involving no drug or device administration.
14. Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 30 days prior to dosing.
15. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
AUC0-240 | Pre-dose, up to Day 57
  Area under the concentration-time curve from time zero to 240hrs
Cmax | Pre-dose, up to Day 57
  The maximal observed concentration
AUC240-672 | Pre-dose, up to Day 57
  Area under the concentration-time curve from time 240 to 672hrs
AUC0-672 | Pre-dose, up to Day 57
  Area under the concentration-time curve from time zero to 672hrs
AUC0-inf | Pre-dose, up to Day 57
  Area under the concentration-time curve from time zero to infinity

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No